CLINICAL TRIAL: NCT03725072
Title: Phase I, Open Label, Single Dose Study to Determine the Pharmacokinetics, Metabolism, and Excretion of [14C]-Evobrutinib in Healthy Participants
Brief Title: Human Absorption, Distribution, Metabolism and Excretion (ADME) of [14C]-Evobrutinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MS200527_0075; 2018-003371-35 (EudraCT Number)
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: [14C]-evobrutinib; Healthy; Pharmacokinetics; Metabolism; Excretion
MeSH Terms: interventions — evobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evobrutinib (Experimental)
  Interventions: Drug: Evobrutinib

INTERVENTIONS:
Drug: Evobrutinib — Participants will receive a single, oral dose of evobrutinib under fasting conditions as a solution, which will contain [14C]-evobrutinib.
  Other Names: M2951

SUMMARY:
The purpose of the study is to determine the absorption, metabolism, and excretion of [14C]-evobrutinib in healthy participants

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring
* Have a body weight within 50.0 to 120.0 kilogram (kg) (inclusive) and body mass index within the range 19.0 - 30.0 kilogram per meter square (kg/m^2) (inclusive)
* Male participants agree to be consistent with local regulations on contraception methods
* Can give signed informed consent
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders
* Prior history of cholecystectomy or splenectomy, and any clinically relevant surgery
* Any surgical or medical condition which might significantly alter the ADME of drugs
* History of any malignancy, chronic or recurrent acute infection
* History of shingles
* History of drug hypersensitivity ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or formulation ingredients
* History of alcoholism or drug abuse
* History of residential exposure to tuberculosis, or a positive QuantiFERON test at screening
* Administration of live vaccines or live-attenuated virus vaccines
* Any condition, including findings in the laboratory tests, medical history, or other screening assessments, that in the opinion of the Investigator constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study's objectives, conduct, or evaluation
* Prior/concomitant therapy
* Relevant radiation exposure
* Clinically relevant findings (excluding minor deviations) in biochemistry, hematology, coagulation and urinalysis
* Vital signs (pulse rate and blood pressure) outside the normal range
* Estimated Glomerular Filtration rate according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
* Semi supine systolic blood pressure (SBP) greater than (>) 140 millimeters of Mercury (mmHg) or less than (<) 90 mmHg, diastolic blood pressure (DBP) > 90 mmHg or < 45 mmHg and pulse rate >= 100 bpm or =< 40 bpm, at admission
* 12-Lead electrocardiogram (ECG) showing a QTcF > 450 millisecond (ms), PR > 215 ms, or QRS > 120 ms
* Positive for hepatitis B surface antigen (HBsAg), hepatitis B core antibody, hepatitis C antibody, or human immunodeficiency virus (HIV) I and II tests at screening
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Total Radioactivity Recovery Rate of Evobrutinib, Total Radioactivity and its Metabolites | Pre-dose up to Day 35 post-dose
Percentage Excretion of Evobrutinib, Total Radioactivity and its Metabolites in Urine and Feces | Pre-dose up to Day 35 post-dose
Renal Clearance of Evobrutinib, Total Radioactivity and its Metabolites | Pre-dose up to Day 35 post-dose
Maximum Observed Plasma Concentration (Cmax) of Total [14C] Radioactivity (Evobrutinib and Metabolites) | Pre-dose up to Day 35 post-dose
Time to Reach Maximum Plasma Concentration (Tmax) of Total [14C] Radioactivity (Evobrutinib and Metabolites) | Pre-dose up to Day 35 post-dose
Terminal Elimination Half-Life (t1/2) of Total [14C] Radioactivity (Evobrutinib and Metabolites) | Pre-dose up to Day 35 post-dose
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Total [14C] Radioactivity (Evobrutinib and Metabolites) | Pre-dose up to Day 35 post-dose
Maximum Observed Plasma Concentration (Cmax) of Evobrutinib | Pre-dose up to Day 35 post-dose
Time to Reach Maximum Plasma Concentration (Tmax) of Evobrutinib | Pre-dose up to Day 35 post-dose
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Evobrutinib | Pre-dose up to Day 35 post-dose
Terminal Elimination Half-Life (t1/2) of Evobrutinib | Pre-dose up to Day 35 post-dose
Apparent Volume of Distribution During Terminal Phase (Vz/f) of Evobrutinib | Pre-dose up to Day 35 post-dose
Apparent Clearance (CL/f) of Evobrutinib | Pre-dose up to Day 35 post-dose

SECONDARY OUTCOMES:
Number of Participants with Clinically Significant Change From Baseline in Vital Signs, Laboratory Parameters and Electrocardiogram Findings | From time of first dose to end of study participation approximately at Day 37
  Number of participants with clinically significant abnormalities will be reported.
Occurrence of Treatment -emergent Adverse Events (TEAEs) and Serious TEAEs | From time of first dose to end of study participation approximately at Day 37
Occurrence of Treatment -emergent Adverse Events (TEAEs) and Serious TEAEs by Severity | From time of first dose to end of study participation approximately at Day 37

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527_0075
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html